CLINICAL TRIAL: NCT07139002
Title: Combined Effect of Sensory Training With Bobath Therapy on Proprioception, Balance, and Motor Function in Patients With Chronic Stroke
Brief Title: Combined Effect of Sensory Training With Bobath Therapy in Patients With Chronic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0281
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Chronic Stroke Patients
Keywords: Bobath Therapy; Sensory training; Chronic Stroke; Balance; Motor function; Proprioception

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bobath Therapy (Other): The group will repeat 10 exercises (facilitated rolling, sitting balance exercises, weight shifting in standing, functional sit-to-stand, stepping practice, reaching activities, wall slides, therapeutic ball exercises, stair climbing practice, and breathing and relaxation techniques) for 8 weeks.
  Interventions: Other: Bobath Therapy
- Sensory Training with Bobath Therapy (Experimental): The group will repeat 9 exercises (texture discrimination, shape, size, and discrimination, tactile recognition, proprioception training, temperature differentiation, tactile localization, sensory mapping, sensory training through functional activities, and tabletop sensory exercises) with Bobath Therapy for 8 weeks.
  Interventions: Other: Bobath Therapy; Other: Sensory Training

INTERVENTIONS:
Other: Bobath Therapy — The group will repeat 10 exercises (facilitated rolling, sitting balance exercises, weight shifting in standing, functional sit-to-stand, stepping practice, reaching activities, wall slides, therapeutic ball exercises, stair climbing practice, and breathing and relaxation techniques) for 8 weeks.
Other: Sensory Training — The group will repeat 9 exercises (texture discrimination, shape, size, and discrimination, tactile recognition, proprioception training, temperature differentiation, tactile localization, sensory mapping, sensory training through functional activities, and tabletop sensory exercises) for 8 weeks.
  Arms: Sensory Training with Bobath Therapy

SUMMARY:
Chronic stroke causes moderate to severe impairments in proprioception, balance, and motor functions, which can impact upon an individual's ability to perform activities of daily living, leading to reduced quality of life and increased dependency. Proprioception, or detecting the body's position in open space, is important for balance and coordinated movement. One therapy uses traditional rehabilitation methods like Bobath theory to increase motor functions, aiming to utilize sensory and movement facilitation. Nonetheless, combining sensory and Bobath therapy could lead to superior outcomes by simultaneously addressing both the proprioceptive deficit and motor skills. The purpose of this project is to explore the combined effect of sensory training and Bobath therapy on proprioception, balance, andmotor function in chronic stroke survivors.

DETAILED DESCRIPTION:
This randomized controlled trial study will take place at Ittefaq (Trust) Hospital, Lahore, with a sample size of 40 participants. Eligible participants will include individuals who are 6 months to 2 years old chronic stroke patients (age group 45 years to 60 years), possess a Mini-Mental State Examination (MMSE) score of 24 or higher, and can provide informed consent. Participants will be selected using nonprobability convenience sampling by using online randomizing tools. The participants will be randomly divided into groups (20 each). The study group will be subjected to combined sensory training and Bobath therapy. The duration of the intervention will be eight weeks, with three sessions per week aimed at improving proprioceptive awareness and motor function. Proprioception will be assessed using the proprioception assessment tool (PAT), joint position sense, and the Romberg test, while balance will be determined using the Berg Balance Scale. The Fugl-Meyer Assessment will be used to measure motor function. The first assessments will be the baseline assessments, done before the intervention, after which a follow-up will be done to measure the efficacy of the combined approach. Statistical analyses will be conducted to assess differences in outcomes between the two groups, helping to determine the effectiveness of combining sensory training with balance and motor function interventions in chronic stroke patients. The findings aim to contribute to the understanding of rehabilitation strategies for this population. Data analysis will be performed by using SPSS 26 software.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female included.
* Age group: 45 years to 60 years.
* Participants diagnosed with chronic stroke 6 months to 2 years.
* Mini-Mental State Examination (MMSE) score of 24 or higher.
* Cannot maintain balance for 30 seconds.
* Ambulate independently for 7 meters.

Exclusion Criteria:

* Participants having conditions other than chronic stroke (Parkinson's disease, Alzheimer's disease, orthopedic pathological condition, etc.).
* Participants having any visual, vestibular, or auditory impairment.
* Participants having any muscular injuries in the previous 6 months.
* Participants with a history of fracture in the previous 6 months.
* Participants with a history of mental illness.
* Participants with cardiovascular complications.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Romberg test | 4 weeks
  Romberg test is popular for assessing proprioception
Joint Position Sense Test | 4 weeks
  Joint Position Sense Test is used for assessing proprioception
Berg Balance scale | 4 weeks
  Berg Balance scale is popular for assessing balance
Timed up and go test | 4 weeks
  Timed up and go test is popular for assessing balance
Fugl-Meyer Assessment Tool | 4 weeks
  Fugl-Meyer Assessment Tool is specific tool that evaluates motor functioning, balance, sensation, and joint functioning in stroke patients

CONTACTS AND LOCATIONS:
Overall Officials: Noshaba Dilshad, MSPT-NM, Principal Investigator — Riphah International University
Locations (1):
- Ittefaq Hospital (Trust), Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No